CLINICAL TRIAL: NCT07284706
Title: Effects of Muscle Warm-Up Phases on Proprioception, Vertical Jump, Agility, and Balance in Professional Youth Soccer Players: A Randomized Study
Brief Title: Warm-Up Phases and Neuromuscular Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Neslihan Altuntas Yilmaz, Assist Prof., Necmettin Erbakan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NEU-PT2025-02; Necmettin Erbakan University (Other: Necmettin Erbakan University)
Record Dates: First submitted 2025-11-27; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Agility; Balance; Warm-up; Proprioception
Keywords: Agility; Balance; Muscle Warm-up; Proprioception; Vertical jump

STUDY DESIGN:
Intervention Model Description: The study included young athletes with at least 3 years of club-level football experience who trained at least 5 days a week for 90 minutes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Program (Experimental)
  Interventions: Other: three warming phases of the muscle

INTERVENTIONS:
Other: three warming phases of the muscle — All assessments will be measured in three warming phases of the muscle. The first phase is the Rest state (Cold state), which is the phase before the training begins. In this phase, the athlete has not warmed up. The second phase is the "Warming state," where the athlete has started the training and has warmed up for 20 minutes. The third phase is the "Post-Training Phase," which occurs 10 minutes after the completion of a 90-minute training session. Measurements will be taken for all three phases.

SUMMARY:
Purpose: This study aimed to examine the effects of different muscle warm-up phases on knee joint proprioception, vertical jump, agility, and balance in professional youth soccer players.

Methods: Twenty-five professional youth football players under 18 were assessed during muscle rest, warm-up, and fatigue phases using tests measuring knee proprioception, dynamic balance, explosive power, and agility.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study was to investigate how different phases of muscle warm-up affect knee joint proprioception, vertical jump performance, agility, and dynamic balance in professional youth soccer players. Understanding these effects is critical for optimizing warm-up protocols to enhance athletic performance and reduce injury risk in this population.

Methods:

Twenty-five male professional youth football players under the age of 18 (mean age 16.5 ± 1.2 years) were randomly selected for this study. Each participant underwent assessments during three distinct muscle states: resting, after warm-up, and post-training fatigue. Knee joint proprioception was evaluated at a 30° angle using a digital inclinometer to measure joint position sense accuracy. Dynamic balance was assessed through the Y-balance test in three directions: anterior, posteromedial, and posterolateral. Explosive power was measured using the Sargent vertical jump test, while agility was tested with the T-test. All measurements were performed in each muscle condition to compare performance across the different warm-up phases.

ELIGIBILITY:
Inclusion Criteria:The study included young athletes with at least 3 years of club-level football experience who trained at least 5 days a week for 90 minutes -

Exclusion Criteria:Individuals with knee pain or a history of knee joint surgery were excluded from this study.

-

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Proprioception Test | It was measured separately in all three phases of exercise. Baseline (resting phase), immediately after the warm-up phase, and immediately after the fatigue phase.
  Knee joint proprioception was assessed using a Baseline Digital Inclinometer (Fabrication Enterprises Inc., USA). Active joint position sense (JPS) of the dominant knee was measured with this device. Participants were seated in a 90° hip and knee flexion position. Initially, the researcher passively positioned the participant's knee at 30° of flexion with eyes open, instructing the participant to memorize the angle. The participant was then asked to close their eyes and actively replicate the target position. The angular deviation from the target was recorded as the proprioceptive error. This procedure was repeated three times, and the mean error was used for analysis .

SECONDARY OUTCOMES:
Sargent Vertical Jump Test | It was measured separately in all three phases of exercise.Baseline (resting phase), immediately after the warm-up phase, and immediately after the fatigue phase.
  The Sargent Jump Test (SJT) was used to evaluate the explosive power of the lower extremities. Participants stood side-on to a wall and extended their dominant arm upward to mark their maximum reach height while standing flat-footed. This point was recorded as the baseline. From a standing position, participants performed a maximal vertical jump and touched the wall at the peak of their jump. The difference between the jump reach and the standing reach height was calculated and recorded as the jump height. Three trials were conducted, and the highest value was used for analysis. A higher score indicates better performance .

OTHER OUTCOMES:
T-Test for Agility | It was measured separately in all three phases of exercise. Baseline (resting phase), immediately after the warm-up phase, and immediately after the fatigue phase.
  Agility was measured using the T-Test, a standardized test involving four cones arranged in a T-shaped configuration. In this setup, three cones were placed in a straight line, each 4.57 meters apart. A fourth cone was placed 9.14 meters perpendicular to the middle cone. Participants were instructed to sprint forward to the center cone, shuffle laterally to each side cone, and then backpedal to the start. The time taken to complete the course was measured using electronic timing gates. Shorter times indicate better agility performance .
Dynamic Balance Test (Y-Balance Test) | It was measured separately in all three phases of exercise. Baseline (resting phase), immediately after the warm-up phase, and immediately after the fatigue phase.
  Dynamic balance was assessed using the Lower Quarter Y-Balance Test. Participants stood barefoot on one leg, placing the stance foot at the center of a Y-shaped grid, with toes behind the starting line. While maintaining single-leg balance, participants reached as far as possible with the non-stance leg in the anterior, posteromedial, and posterolateral directions without losing balance or touching down. Each participant performed three trials per direction, and the average reach distance was calculated for each. Higher reach distances indicate better dynamic balance performance .

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Altuntaş YILMAZ, Assistant Professor, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Nezahat Keleşoğlu Faculty of Health Sciences, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The primary reasons why Individual Participant Data (IPD) cannot or may not be shared stem from Ethical Review Board (IRB/IEC) decisions and legal obligations regarding participant privacy.

REFERENCES:
- [Background] 12. Davis DS, Briscoe DA, Markowski CT, Saville SE, Taylor CJ. Physical characteristics that predict vertical jump performance in recreational male athletes. Phys Ther Sport. 2003;4(4):167-74